CLINICAL TRIAL: NCT00635869
Title: Advancing Research and Clinical Practice Through Close Collaboration (ARCC): A Pilot Test of an Intervention to Improve Evidence-Based Care and Patient Outcomes
Status: Completed | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Priscilla Sandford Worral, Coordinator of Nursing Research, University Hospital, SUNY Upstate Medical University
Other Study IDs: 5199
Record Dates: First submitted 2008-03-07; First posted 2008-03-14 (Estimated); Last update posted 2008-03-14 (Estimated); Status verified 2008-03

CONDITIONS: Evidence-Based Medicine; Physician-Nurse Relations
Keywords: evidence based practice beliefs; evidence based practice implementation; evidence based practice knowledge; nurse physician collaboration

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- ARCC standard: RNs on unit receiving basic ARCC information with staff nurse champion
  Interventions: Behavioral: ARCC standard information
- ARCC enhanced: RNs on unit receiving ARCC standard content plus with an EBP mentor
  Interventions: Behavioral: ARCC enhanced
- C: RNs on the unit receiving the placebo intervention
  Interventions: Behavioral: Placebo

INTERVENTIONS:
Behavioral: ARCC standard information — EBP didactic education sessions, EBP toolkit, environmental prompts, identification of an EBP champion among unit staff RNs
  Groups: ARCC standard
Behavioral: ARCC enhanced — same as ARCC standard plus EBP mentor on-site twice each week plus available by e-mail for consultation
  Groups: ARCC enhanced
Behavioral: Placebo — didactic education sessions on physical assessment
  Groups: C

SUMMARY:
The primary aim of this pilot study is to evaluate the effects of two variations of the ARCC Intervention Program on nursing processes and outcomes (job satisfaction, group cohesion, EBP knowledge, EBP implementation, EBP beliefs), patient/family outcomes (e.g. pt/family satisfaction with care), and institutional processes and outcomes (e.g. nurse-physician collaboration, cost, RN turnover, incidence frequency relevant to the topic). Secondary aims are to test the feasibility of study methods and reliability and validity of questionnaires.

This study is designed as a three-group randomized clinical trial with repeated measures. Three inpatient units (medicine, surgery, surgical intensive care) will be randomly assigned to one of three interventions: ARCC enhanced (didactic content presentations, use of an EBP tool kit which will stay on the unit, environmental EBP prompts, availability of an EBP coach on the unit); ARCC standard (all of the above, but without the coach); non-EBP intervention (didactic content and environmental prompts, but not related to EBP; placebo). The interventions will be implemented over an estimated 14 weeks, including a 4-week training period, and an estimated 10 weeks to implement an EBP initiative that the nurses on the two ARCC intervention units will develop.

Baseline information and questionnaires will be collected from nurses at the start of the study, and again at completion of the intervention phase. Outcome data will be collected from nurses approximately 10 weeks after implementation of the ARCC interventions are completed (i.e., 22 weeks after the study is commenced). Nurse-physician collaboration data will be collected from physicians working with study unit nurses as well as from the nurses. Patient satisfaction data will not be separately collected in this study, but will include use of unit-level Press-Ganey scores immediately prior to and over the study time period. Unit level and institutional RN turnover will be tracked monthly during the entire study period and will be compared across units at the same time as well as compared within each study over time (i.e., unit retention during those same months in the previous year). Costs of each EBP intervention will be tracked during the study and compared descriptively. Survey data will be analyzed using analysis of variance statistics. Questionnaires will be tested for reliability and construct validity. Because this is a pilot study, statistically significant differences are not expected, however, effect sizes will be calculated

ELIGIBILITY:
Inclusion Criteria:

* employed by Upstate
* working full or part time on study unit
* able to attend all education sessions

Exclusion Criteria:

* employed by temporary agency
* not able to attend all education sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Registered Nurse staff working on inpatient study units (medicine, surgery, surgical intensive care)
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2005-09; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
EBP beliefs | baseline, week 5, week 16, week 24

SECONDARY OUTCOMES:
EBP Implementation | baseline, week 5, week 16, week 24

CONTACTS AND LOCATIONS:
Overall Officials: Priscilla S Worral, PhD, RN, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- University Hospital, SUNY Upstate Medical University, Syracuse, New York, United States